CLINICAL TRIAL: NCT03364023
Title: Post-Market Registry Of Stroke Patients Treated With Medtronic Neuro Thrombectomy Devices to Collect Real World Data in South East Asia (PROSPR-SEA)
Brief Title: Post-Market Registry Of Stroke Patients Treated With Medtronic Neuro Thrombectomy Devices to Collect Real World Data in South East Asia
Acronym: PROSPR-SEA
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16066SOLSEA
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Acute Ischemic Stroke Patients: Acute Ischemic Stroke (AIS) patients treated with Medtronic Market-Released Neurothrombectomy Device
  Interventions: Device: Neurothrombectomy

INTERVENTIONS:
Device: Neurothrombectomy — Medtronic Market-Released Neurothrombectomy Device

SUMMARY:
The purpose of this post-market registry is to collect real-world data associated with the use of Medtronic market-released neurothrombectomy devices in acute ischemic stroke (AIS) patients from countries in South East Asia.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry designed to collect real world data associated with the use of Medtronic market-released neurothrombectomy devices in acute ischemic stroke (AIS) patients from countries in South East Asia, including Singapore, Thailand and Vietnam. The primary objective of this registry is to assess clinical outcomes associated with the use of these devices in patients experiencing AIS due to large intracranial vessel occlusion within 8 hours of symptom onset. This registry may enroll up to 500 patients.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402 (j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402 (j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

1. Subject/subject's legally authorized representative has given Informed Consent according to country regulations, and/or EC requirements.
2. Subject has experienced an Acute Ischemic Stroke due to large intracranial vessel occlusion in at least one of the following intracranial vessels: internal carotid artery (ICA), M1 and M2 segments of the middle cerebral artery (MCA), basilar, and vertebral arteries.
3. Subject has been or will be treated with a Medtronic market-released neurothrombectomy device as the initial device used to remove the thrombus.
4. Subject is willing to participate in a 90-day follow-up visit.
5. Treatment within 8 hours of stroke symptom onset (defined as stroke onset to access puncture).

Exclusion Criteria:

1. Concurrent participation in another mechanical neurothrombectomy device trial or any other clinical trial with an active treatment arm or where the study procedure or treatment might confound the study analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AIS patients treated with a Medtronic market-released neurothrombectomy device.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ka Sing Lawrence Wong, MD, Principal Investigator — Chinese University of Hong Kong
Locations (10):
- Singapore (3):
  - National Neuroscience Institute, Singapore
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Thailand (3):
  - Prasat Neurology Institute, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Vietnam (4):
  - 108 Military Central Hospital, Hanoi
  - Bach Mai Hospital, Hanoi
  - Ho Chi Minh City Medicine and Pharmacy University, Ho Chi Minh City
  - The People's 115 Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Ischemic Stroke Patients: Acute Ischemic Stroke (AIS) patients treated with Medtronic Market-Released Neurothrombectomy Device due to large intracranial vessel occlusion within 8 hours of symptom onset.
Period: Overall Study
Arm/Group | Acute Ischemic Stroke Patients
Started | 183
Completed | 166
Not Completed | 17
Not completed — Lost to Follow-up | 3
Not completed — Death | 14

BASELINE CHARACTERISTICS:
Arm/Group | Acute Ischemic Stroke Patients
Number analyzed (Participants) | 183
Age, Continuous [Median (Standard Deviation); unit: Years] | 64.89 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.13 (3.91)
Pre-stroke mRS [Count of Participants; unit: Participants] — The modified Rankin Scale (mRS) measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale ranges from 0-6, with lower values representing a better outcome.
  0-No symptoms at all
  1. No significant disability despite symptoms
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 3 Moderate disability; requiring some help 4 Moderately severe disability 5 Severe disability; bedridden, incontinent and requiring constant nursing care and attention 6 Dead
  Participants
    mRS = 0 | 147
    mRS = 1 | 14
    mRS = 2 | 2
    mRS = 3 | 2
    mRS = 4 | 2
    mRS = 5 | 1
    Not Done | 15
Baseline NIHSS [Mean (Standard Deviation); unit: units on a scale] — The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
  units on a scale | 15.20 (5.88)

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale (mRS) at 90 Days
Description: mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 90 Days Post Procedure
Measure: Number; unit: Participants
Arm/Group | Acute Ischemic Stroke Patients
Number analyzed (Participants) | 180
Participants
  mRS = 0-2 | 112
  mRS = 3-6 | 68

2. Secondary Outcome: Number of Participants With Symptomatic Intracranial Hemorrhage (sICH) at 24 Hrs ± 8 Hrs Post Procedure
Description: Number of participants with symptomatic Intracranial hemorrhage (sICH) is defined as >/= 4 points worsening from baseline on the National Institutes of Health Stroke Scale (NIHSS) associated with an image finding of intra-cranial hemorrhage (i.e., intracerebral or intraventricular) at 24 +/- 8 hrs post procedure.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
Time Frame: 24 hrs ± 8 hrs post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Ischemic Stroke Patients
Number analyzed (Participants) | 183
Participants | 14

3. Secondary Outcome: All-Cause Mortality Through 90 Days Post Procedure
Description: Death through 90 days post procedure classified as neurological or non-neurological, with event leading to death.
Time Frame: 90 Days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Ischemic Stroke Patients
Number analyzed (Participants) | 183
Participants | 14

4. Secondary Outcome: Incidence of Emboli in New Territory (ENT) at 24 Hrs ± 8 Hrs Post Procedure
Description: Emboli in New Territory (ENT) is defined as embolization territories outside of the target downstream territory.
Time Frame: 24 hrs ± 8 hrs post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Ischemic Stroke Patients
Number analyzed (Participants) | 183
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the point of consent through 90 day follow up visit.
Description: For the purpose of this real-world registry, only the following Serious Adverse Events were collected:
  * Symptomatic Intracranial Hemorrhage (sICH) at 24 ± 8 hrs post procedure
  * Death through 90 days post procedure classified as neurological or non-neurological, with event leading to death
  Other [Not including Serious] Adverse Events were not monitored/assessed for this registry.
Arm/Group | Acute Ischemic Stroke Patients
All-Cause Mortality (participants affected / at risk) | 14/183
Serious Adverse Events (participants affected / at risk) | 14/183
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Ischemic Stroke Patients (N=183)
Symptomatic Intracranial Hemorrhage (sICH) (Nervous system disorders) | 14 — Symptomatic Intracranial Hemorrhage (sICH) at 24 ± 8 hrs post procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03364023/Prot_SAP_000.pdf